CLINICAL TRIAL: NCT03600662
Title: TriRec - Trileaflet Reconstruction of the Aortic Valve
Brief Title: TriRec - Trileaflet Reconstruction of the Aortic Valve With Autologous Pericardium
Acronym: TriRec
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Department of Cardiovascular Surgery, German Heart Center Munich (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 389/17S
Record Dates: First submitted 2018-05-30; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Alternative Surgical Treatment for Aortic Valve Disease
Keywords: aortic stenosis; aortic regurgitation; Trileaflet reconstruction of the aortic valve; Biological aortic valve prosthesis; Effective orifice area
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TriRec (Experimental): Trileaflet Reconstruction of the Aortic Valve
  Interventions: Other: TriRec
- Aortic valve replacement (Experimental): Biological prosthesis, Device: St. Jude Medical Trifecta GT
  Interventions: Other: Aortic valve replacement

INTERVENTIONS:
Other: TriRec — Trileaflet Reconstruction of the Aortic Valve
  Arms: TriRec
Other: Aortic valve replacement — Biological Prosthesis, Device: St. Jude Medical Trifecta GT
  Arms: Aortic valve replacement

SUMMARY:
Reconstruction of the aortic valve using the tri-leaflet repair technique is non-inferior with regard to effective orifice area (EOA) to surgical aortic valve replacement (SAVR) with a biological prosthesis (St. Jude Trifecta GT) as gold- standard.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 50 years
* Documented symptomatic moderate or greater aortic stenosis or severe insufficiency
* Aortic annulus > 19 mm
* Written informed consent of the patient.

Exclusion Criteria:

* Concomitant intervention of the aortic root
* Concomitant intervention of the aortic arch
* Concomitant valve surgery
* Emergency surgery for any reason
* Neurological events (i.e. stroke, TIA) within 6 months preoperatively
* Coagulation disorders (including thrombocytopenia < 100.000/ml)
* Porcelain aorta
* Active endocarditis or other active systemic infections
* Participating in another trial that may influence the outcome of this trial
* Pregnancy
* Dual antiplatelet therapy
* Previous cardiac surgery (excluding percutaneous procedures)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Effective orifice area | 10th postoperative day +/- 4 days
  Effective orifice area in cm2 (EOA) either after the TriRec- procedure or surgical valve replacement with the St. Jude Medical Trifecta GT Valve, measured by echocardiography

SECONDARY OUTCOMES:
Effective orifice area | after 6 months, 1 year and thereafter annually until the 10th postoperative year
  Effective orifice area in cm2 (EOA) either after the TriRec- procedure or surgical valve replacement with the St. Jude Medical Trifecta GT Valve, measured by echocardiography
Maximum and mean aortic pressure gradients | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Estimation of aortic regurgitation, if applicable | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Left ventricular ejection fraction | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Left ventricular endsystolic and -diastolic diameter | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Left ventricular endsystolic and -diastolic volume | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Left atrial diameter | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Freedom from aortic valve reintervention at discharge | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year
Freedom from Mortality | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Freedom from Stroke | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Freedom from Myocardial infarction | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Freedom from conduction disturbances leading to permanent pacemaker implantation | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Freedom from Endocarditis | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.
Freedom from Bleeding requiring re-thoracotomy | 10th postoperative day +/- 4 days, after 6 months, 1 year and thereafter annually until the 10th postoperative year.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Krane, MD, PhD, Study Chair — Department of Cardiovascular Surgery, German Heart Center Munich
Locations (1):
- Department of Cardiovascular Surgery, German Heart Center Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No